CLINICAL TRIAL: NCT03937167
Title: Benefits of a Psychotherapy Group Program as Oppossed to the Standard Method in the Treatment of Obesity. A Randomized Controlled Trial.
Brief Title: Benefits of Group Psychotherapy Programs in the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Infanta Leonor (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Javier Quintero, Psychiatry Department Head, Hospital Universitario Infanta Leonor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PsicoObe
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Psychotherapy; Psychotherapy, Group
Keywords: obesity; Psychotherapy; Psychotherapy Group
MeSH Terms: conditions — Obesity | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard treatment at Hospital Infanta Leonor with Endocrinology and Psyquiatry
- Completers (Experimental): Randomized to treatment AND complete treatment 14 sessions are needed
  Interventions: Other: Psychotherapy group
- Drop-out (No Intervention): Randomized to treatment BUT do not assist or do not complete treatment Less than 14 sessions

INTERVENTIONS:
Other: Psychotherapy group — Added to standard treatment patients will participate in a standardized group of psychological intervention. 21 sessions with 10 to 12 members closed-ended groups.
  Arms: Completers

SUMMARY:
Obesity has reached pandemic proportions in recent years, affecting not only the physical health, but also the mental health, of obese people. According to Spain's National Health Survey 2011-12, the prevalence of obesity in the adult population of Spain was 17%, having increased by 2.5% since 2006. Therefore, a constant and worrying increase in the prevalence of obesity is being observed, which is having a great impact, both individually, in terms of health and quality of life, and socially, inter alia, by raising health expenditure due to increased morbidity.

In this context, the desirability of a comprehensive approach that includes psychological intervention in attending obese patients (Rev Cochrane, 2006), has been given greater prominence. Paying attention to the emotional and psychopathological aspects related to obesity has proven to be an action that could have positive impact on obesity intervention models.

The aim of this project is to measure, through a clinical trial, the efficacy of a psychotherapy group program for obesity patients who are attended by the consulting endocrinologist at the Infanta Leonor Hospital (Madrid). The impact of body mass index, psychological wellbeing, psychopathology and quality of life of two experimental study groups will be compared, one a control group of patients that follows the standard treatment, the other an experimental group that follows not only the standard treatment, but also the psychotherapy group intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 and younger than 65.
* Body mass index of 30 or higher.
* Candidate to a specific obesity treatment.
* Accept psychological attention.
* Able to understand and consent participation.
* Able to speak, write and read in Spanish.
* Committed to assist weekly for 6 months

Non-inclusion Criteria:

* Obesity related to a non- stabilized hormonal disorder.
* Severe mental disorders requiring specific treatment resources.
* Cognitive or sensitive deficits.
* Having had bariatric surgery within last 2 years.

Exclusion criteria:

* Pregnancy during treatment
* Bariatric surgery during treatment
* Addictive disorder as a principal diagnosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
weight difference | 1 year
  Difference between the initial and final weight in kilograms

SECONDARY OUTCOMES:
Global Severity Index (GSI) | 1 year
  Global psychopathology measured by Symptom Checklist-90-Revised (SCL-90-R). T score.
Positive Symptom Distress Index (PSDI) | 1 year
  Style of response to distress measured by Symptom Checklist-90-Revised (SCL-90-R). T score.
Positive Symptom Total (PST). | 1 year
  count of all the items with non-zero responses at Symptom Checklist-90-Revised (SCL-90-R). T score.
Eating disorder risk (EDRC) | 1 Year
  disfunctional eating behavior assessed by Eating Disorders Inventory 3rd Edition (EDI-3). T score. It is an index calculated by combining 3 scales: drive for thinness, body dissatisfaction, and bulimia
Physical quality of life | 1 year
  perceived physical quality of life assessed by Quality of Life Cuestionnaire SF-36
Mental quality of life | 1 year
  perceived mental or psychic quality of life assessed by Quality of Life Cuestionnaire SF-36
Mediterranean Diet Adherence | 1 year
  Mediterranean Diet Adherence measured by Test KIDMED
Motivation to change | 1 year
  Motivation to change assessed by University of Rhode Island Change Assessment (URICA). 4 scales are measured: precontemplation, contemplation, action and maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Félix, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No